CLINICAL TRIAL: NCT06193642
Title: Increasing Knowledge on Osteogenesis Imperfecta by Collecting and Integrating Epidemiological Data, Genetic Information, and Functional Performance From Movement Analysis
Brief Title: Increasing Knowledge on Osteogenesis Imperfecta by Collecting Epidemiological Data
Acronym: 4FRAILTY
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 4FRAILTY
Record Dates: First submitted 2023-11-23; First posted 2024-01-05 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-03

CONDITIONS: Osteogenesis Imperfecta
MeSH Terms: conditions — Osteogenesis Imperfecta

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental (Experimental): Through gait analysis acquisition sessions in the most comprehensive configuration possible on a test group of patients, the aim is to identify measures to be collected at regime for simplified evaluation including patient acceptability.
  Patients will be asked to complete quality of life questionnaires.
  Interventions: Other: experimental

INTERVENTIONS:
Other: experimental — Subjects diagnosed with OI will undergo a series of assessments using sensor imaging and Gait-Analysis; we will proceed with a careful and detailed collection, analysis and evaluation of functional data typical of Gait-Analysis studies, aimed at identifying that subset of parameters that will prove most interesting and useful for the purposes of the study, thus identifying the sensors and algorithms that can precisely produce the most usable synthetic information for defining the quality of motor function in these patients.

SUMMARY:
interventional pilot study with the enrollment of patients affected by Osteogenesis Imperfecta

DETAILED DESCRIPTION:
Subjects diagnosed with Osteogenesis Imperfecta will be undergoing, after collection of informed consent, to a series of assessments using sensor imaging and Gait-Analysis and collection of specific parameters

ELIGIBILITY:
Inclusion Criteria:

* Patients with Osteogenesis Imperfecta (clinical diagnosis) able to perform the gait-analysis movement data acquisition session, in the most complete instrumental configuration, i.e., with kinematics, dynamics and electromyography; it will naturally be evaluated which motor tasks are safely executable and which are not.
* All patients of both sexes will be included
* Patients in the age range: 8-60 will be included

Exclusion Criteria:

* Subjects who do not fit the inclusion criteria

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2023-01-20 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-11-30 (Estimated)

PRIMARY OUTCOMES:
Gait-Analysis | through study completion, an average of 1 year
  Parameter detection via specific sensors including Inertial Motion Units

SECONDARY OUTCOMES:
quality of life questionnaires | through study completion, an average of 1 year
  quality of life assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

REFERENCES:
- [Result] Colnaghi S, Rezzani C, Gnesi M, Manfrin M, Quaglieri S, Nuti D, Mandala M, Monti MC, Versino M. Validation of the Italian Version of the Dizziness Handicap Inventory, the Situational Vertigo Questionnaire, and the Activity-Specific Balance Confidence Scale for Peripheral and Central Vestibular Symptoms. Front Neurol. 2017 Oct 10;8:528. doi: 10.3389/fneur.2017.00528. eCollection 2017. PMID 29066999
- [Result] Benedetti MG, Catani F, Leardini A, Pignotti E, Giannini S. Data management in gait analysis for clinical applications. Clin Biomech (Bristol). 1998 Apr;13(3):204-215. doi: 10.1016/s0268-0033(97)00041-7. PMID 11415789